CLINICAL TRIAL: NCT02927886
Title: Per-oral Endoscopy Pyloromyotomy (G-POEM) in the Treatment of Refractory Diabetic Gastroparesis : Prospective Evaluation of Efficacy
Acronym: G-POEM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-17; 2016-A01365-46 (Other: ANSM)
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Pyloromyotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Per-oral Endoscopy Pyloromyotomy (G-POEM) (Experimental)
  Interventions: Procedure: Per-oral endoscopy pyloromyotomy
- Intrapyloric injection of botulinum toxin (Placebo Comparator)
  Interventions: Procedure: Intrapyloric injection of Botulinum toxin

INTERVENTIONS:
Procedure: Per-oral endoscopy pyloromyotomy
  Other Names: G-POEM
  Arms: Per-oral Endoscopy Pyloromyotomy (G-POEM)
Procedure: Intrapyloric injection of Botulinum toxin
  Arms: Intrapyloric injection of botulinum toxin

SUMMARY:
The objective of the study is to document the clinical efficacy and complications of endoscopic pyloromyotomy in patients with refractory gastroparesis (diabetic, post-operative and idiopathic), compared to Botulinic toxin injection intra-pyloric the results of which are close to the placebo.

DETAILED DESCRIPTION:
Gastroparesis is a functional disease affecting 4% of the population, which is consecutive to diabetes in 30% of cases and considerably alters the patients' quality of life. The diagnosis is based on gastric fullness symptoms, endoscopy and gastric emptying scintigraphy. The therapeutic alternatives including drug therapies (Metoclopramide, Erythrocin), surgery (Electric gastric stimulation) or endoscopy (Botulinic toxin), are insufficiently effective. Two surgical series suggested an interesting efficacy of laparoscopic pyloroplasty, which remains invasive for a motility disorder. More recently, an US team performed the first case of G-POEM with an excellent outcome and no adverse event. This promising result was confirmed by a Brazilian case, a short retrospective series (7 patients) and the first European case performed and published by our team that has performed 5 cases since. Based on experience, it is proposed a prospective monocentric study to evaluate the efficacy of the G-POEM technique on refractory gastroparesis. This study will include 40 patients on a period of three years, whom suffer from refractory gastroparesis, confirmed by clinical evaluation (GCSI and analogic visual scale), upper GI endoscopy and gastric emptying scintigraphy at the inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years.
* Presenting a clinical refractory gastroparesis for> 1 year, that is to say whose functional nonspecific symptoms persisting despite medical therapy (prokinetic) optimal.
* Having a calculation before inclusion GCSI score (Gastroparesis Cardinal Symptom Index) and a scan of the pathological gastric emptying finding gastroparesis older than 3 months.
* No history of gastric surgery (partial gastrectomy Sleeve gastrectomy, ...) or esophageal surgery
* Not having endoscopic gastric lesions (ulcers antro-pyloric cancer).
* Having no indication against anesthetic.
* Having consented to participate in the study.
* Affiliated with a social security scheme (beneficiary or assignee).

Exclusion criteria:

* Minors.
* Pregnant or breastfeeding
* Having an anesthetic against indication.
* Scan the normal gastric emptying
* Under curative dose anticoagulants whose suspension is inappropriate.
* Under dual anti-platelet aggregation whose suspension is inappropriate.
* Being unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-09 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Gastroparesis Cardinal Symptom Index score calculation | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Geindre, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Gastro-entérologie, Hôpital Nord ,Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No